CLINICAL TRIAL: NCT03951337
Title: Evaluation of 64Cu-ATSM PET/CT in Predicting Neo Adjuvant Treatment Response in Locally Advanced Rectum Cancer
Brief Title: 64Cu-ATSM PET/CT in Rectum Cancer (TEP 64Cu-ATSM-Rectum)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Fondation ARC (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ICO-N-2017-14
Record Dates: First submitted 2019-04-26; First posted 2019-05-15 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Rectal Cancer
Keywords: 64Cu-ATSM; neoadjuvant treatment; chemoradiotherapy; surgery; Positron Emission Tomography (PET)/CT scan; Prediction of response to treatment; Rodel score
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Multicentric, open prospective study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 64Cu ATSM (Experimental): pretherapeutic 64Cu-ATSM PET/CT scan
  Interventions: Drug: 64Cu-ATSM

INTERVENTIONS:
Drug: 64Cu-ATSM — 64 Cu-ATSM PET/CT scan

SUMMARY:
This phase II trial is assessing how 64Cu-ATSM (64Cu-copper(II) diacetylbis(N4-methylthiosemicarbazone)) PET/CT scan could predict neo adjuvant treatment response in rectum cancer locally advanced

DETAILED DESCRIPTION:
The purpose of this study is to evaluate early and late tumor uptake of 64Cu-ATSM in predicting histological response to neo-adjuvant chemo-radiotherapy treatment in patients with locally advanced rectal cancer.

Patients receive pre-therapeutic CT scan, Pelvic MRI and 18FDG (fluorodeoxyglucose) PET/CT (positron emission tomography) scan within 45 days before enrollment.

64Cu-ATSM PET/CT scan is done before chemoradiotherapy treatment start. About 3 MBq/Kg of 64Cu-ATSM are injected intravenously, two acquisition sequences are performed 1 hour and 23 to 25 hours after injection in order to evaluate early and late tumor uptake of 64Cu-ATSM.

Patients are treated for 5 weeks by Capecitabine chemotherapy (1600 mg/m2/day) combined to 50 Gy radiotherapy.

Pelvic MRI is performed 4 weeks after chemotherapy in order to evaluate the treatment efficacy.

Surgery is scheduled 6 to 8 weeks after chemoradiotherapy. Tissue samples from previously collected rectal biopsy (obtained for diagnosis) and from surgery are used for assessing oxidative stress markers by Immuno-histochemical analysis.

Chest, abdomen and pelvis CT scan is performed every 6 months after surgery in order to assess progression free survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectum adenocarcinoma
* Locally advanced, non metastatic disease, with or without locoregional lymph node involvement (greater than or equal to T3 +/- N), first-line therapy
* 18 Years and older
* Performance Status equal to 0 or 1
* Fertile patients must use effective contraception
* Hemoglobin greater than 9g/dl, neutrophils greater than 1 500/mm3, platelets greater than 100 000/mm3
* Creatinine clearance greater than or equal to 50ml/min
* Plan to receive treatment with concurrent chemotherapy and radiation therapy followed by surgery
* Totality of the tumor included in the radiotherapy field
* Written informed consent
* Patient must be affiliated to a Social Health Insurance

Exclusion Criteria:

* metastatic disease
* Patient contraindicated for capecitabine or 5FU (5-Fluoro-Uracile) derivatives (history of severe and unexpected reactions to fluoropyrimidine-containing therapy, known hypersensitivity to 5FU, to any of the excipients, or known total DPD (dihydropyrimidine déshydrogénase) deficiency)
* Known Contraindication to perform MRI
* Previous treatment with pelvic radiotherapy
* Chronic inflammatory bowel disease, malabsorption, lack of colonic integrity
* Diarrhea grade greater than 2
* Contraindication to surgery
* Bilateral total hip prosthesis
* Other malignancy treated within the last 5 years (except non-melanoma skin cancer or in situ carcinoma of the cervix)
* Pregnant or nursing patient
* Individual deprived of liberty or placed under the authority of a tutor
* Impossibility to submit to the medical follow-up of this clinical trial for geographical, social or psychological reasons
* Agitation; impossibility of lying motionless for at least 1 hour, or known claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2019-04-26 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Relationship between early tumor uptake of 64Cu-ATSM PET/CT images and prediction of histological response to neo-adjuvant chemo-radiotherapy treatment | 4 months
  Early tumor uptake of 64Cu-ATSM will be assessed by SUV (Standardized Uptake Value) measurement, histological response Will be assessed by Rodel grading (Tumor Regression Grading)

SECONDARY OUTCOMES:
Relationship between late tumor uptake of 64Cu-ATSM PET/CT images and prediction of histological response to neo-adjuvant chemo-radiotherapy treatment | 4 months
  Late tumor uptake of 64Cu-ATSM will be assessed by SUV (Standardized Uptake Value) measurement, histological response Will be assessed by Rodel grading (Tumor Regression Grading)
Correlation between 64Cu-ATSM uptake and oxidative stress markers | 4 months
  Aggressive zones corresponding to high redox potential areas will be assessed by Immuno-histochemical analysis on the surgical sample and on the pre-therapeutic biopsy
Progression free survival | 2 years
  Progression Free survival is the delay between surgery and the date of documented disease progression
18FDG-PET/CT and 64Cu-PET/CT uptakes | 45 days
  Correlation between 18FDG-PET/CT and 64Cu-PET/CT uptakes
Comparison between early and late 64Cu-ATSM uptakes in 64Cu-ATSM PET/CT images | 45 days
  Early and Late tumor uptake of 64Cu-ATSM will be assessed by SUV (Standardized Uptake Value) measurement
64Cu-ATSM toxicity | 45 days
  64Cu-ATSM toxicity will be assessed by vital signs monitoring within 2 hours after 64Cu-ATSM injection

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde COLOMBIE, MD, Principal Investigator — Institut de Cancerologie de l'Ouest
Locations (5):
- France (5):
  - Institut de Cancerologie de l'Ouest (ICO), Angers
  - CHU de BREST, Brest
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut de cancerologie de l'Ouest, Saint-Herblain